CLINICAL TRIAL: NCT00174876
Title: An Open-Label Study of Aripiprazole (Abilify) as an Augmentation Agent in Patients With Treatment-Resistant Depression
Brief Title: Aripiprazole as Augmentation for TRD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4894; 1040272-1 32678
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-09-18 (Estimated); Status verified 2008-09

CONDITIONS: Depression
Keywords: depression
MeSH Terms: conditions — Depression

INTERVENTIONS:
Drug: Drug Abilify

SUMMARY:
A sizeable minority of patients suffering from major depression do not have their full set of depressive symptoms relieved by a single medication. Often times, a second medication is added to a patient's first antidepressant to obtain a better response in hopes of getting the depressed patient into full remission from symptoms.

A typical psychiatric approach of recent has been to add one of the newer anti-schizophrenia medications to an existing FDA approved antidepressant in order to achieve better serotonin levels in the depressed patient's brain. This optimization of brain serotonin helps to alleviate more depressive symptoms. The newest antipsychotic medication to be FDA approved is Aripiprazole (Abilify). It may be particularly effective as it may safely elevate sertotonin through receptor 1a stimulation, receptor 2a blockade. It may also facilitate low levels of dopamine transmission which is truly novel for this agent when compared to other schizophrenia drugs. Depressed patients also tend to lack dopamine in their brains. This makes Aripiprazole and ideal agent to boost both serotonin and dopamine simultaneously. In theory, this may be an effective way to alleviate more depressive symptoms.

The author suggests to enroll 10 subjects initially in open label fashion to take Aripiprazole plus their current FDA approved antidepressant to see if further elimination of depressive symptoms occurs and to show this pharmacological approach as a tolerable combination of medications. If there are no major safety issues, an amendment to allow 10 additional subjects will be forwarded to provide a better tolerability sample size.

DETAILED DESCRIPTION:
This is a prospective, open-label study that will examine the clinical utility and safety of adding the atypical antipsychotic aripiprazole as an augmenting agent to antidepressant therapy in treatment-resistant depressed patients. The author's a priori hypothesis is that aripiprazole plus a current FDA approved antidepressant will result in significant reductions in depressive symptoms over 6 weeks. Responders (>50% improvement in baseline HAM-D score) will be asked to voluntarily continue in a 6 week open-label extension in order to show that antidepressant effects of aripiprazole are longstanding in nature.

After screening and consenting and liaison with a primary prescriber, 10 eligible subjects will receive aripiprazole 10-30 mg per day as an augmentation agent in combination with their current FDA approved antidepressant medication. The dose of the subject's original antidepressant will remain unchanged during the study unless subject notes intolerable newly emergent antidepressant-related side effects. Based on tolerability and response, aripiprazole will be started at 5 mg per day and augmented as follows (baseline, end of week 1, end of week 2, end of week 4, and termination visit end of week 6) at 5 mg per day increments, the maximum dose being 30 mg per day for patients who are taking antidepressants that have no pre-existing significant inhibitory effect on CYP450 2D6 enzyme system. However, if the patient is taking any antidepressant that has significant CYP450 2D6 enzyme inhibitory properties, that may affect the metabolism of aripiprazole (e.g. paroxetine, fluoxetine), the maximum dose will be 15 mg per day (50% less than the maximum recommended dose). These dose ranges have been chosen because they capture the mean effective dose for ameliorating depressive symptoms in schizophrenia. The dose will be titrated upward or downward based on clinical response. Other psychotropic medications will be permitted during the study if deemed necessary to control side effects (hypnotics, anxiolytics, antimuscarinics, beta blockers, etc.). Subjects who have been on a stable dose of hypnotic or anxiolytic (GABA or Histamine-based) for at least 4 weeks prior to study entry may opt to continue these at current dose or be washed out prior to study start. Aripiprazole will be dispensed biweekly and the participants will be followed for 6-weeks. Participants will be monitored every other week by the HAMD (blinded), CGI, and SAFTEE. Vital signs and weight will also be taken at each visit. After 6 weeks, there will be a two-week taper of aripiprazole (50% reduction in dose per week). Compliance will be measured by pill count All subjects will be voluntarily offered to stay in the study for an additional six weeks where they will meet one final time at the end of week 12 to re-evaluate safety and effectiveness of longer term aripiprazole augmentation. Subjects would then go through a two week taper as above. Subjects who do not wish to continue an additional six weeks may opt out of the study at the original 6 week termination mark. If interim safety analysis (by independent psychiatrist TBD) suggests good safety profile and amendment will be sent to the IRB asking for 10 additional subjects to be enrolled.

Primary and secondary measures and safety evaluations: The primary measures of the study will be changes in HAMD scores over time (we will monitor this to make sure depression scores do not worsen with aripiprazole); the secondary efficacy measure will be changes in CGI scores over time. Safety evaluations will be determined by the SAFTEE rating scale and patient AE reports. An Expectancy Scale will be given to determine if subjects' level of perceived confidence in the drug correlates to the outcomes noted above. This is a superficial way to look at placebo-like rates when placebo is not used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria: males or females age 18 to 65 years, DSM-IV episode of Major Depression non-psychotic, ≥14 score on the 17-item HRSD, adequate trial with two antidepressants (see definition above of 'adequate trial'), ability to receive and give informed consent, if patients are of child-bearing potential (male or female), use of an effective contraceptive is required for at least one month prior to the screening Visit and documentation of a negative pregnancy (female) test upon entry into the study.

Exclusion Criteria:

* Exclusion Criteria: bipolar or psychotic depression, overt personality disorder, currently suicidal or a history of suicide attempt in the previous 6 months, current substance abuse or history of substance abuse in the previous 12 months, history of hypersensitivity to aripiprazole, treatment with antipsychotic medications in the previous 3 months, serious or unstable medical disorders which in and amongst themselves may lend to morbidity or mortality during study, any medical illness with relative contraindication for aripiprazole use, starting or terminating psychotherapy during the previous 12 weeks, ECT treatment in the previous 3 months, pregnancy or planning pregnancy, history of severe head injury with sequelae, comorbid anxiety condition which has been focus of clinical attention in previous 6 months (remitted GAD, OCD, Panic, Social Anxiety, PTSD may be allowed).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-07; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L. Schwartz, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States